CLINICAL TRIAL: NCT05294926
Title: Comparison Of Deep Versus Moderate Neuromuscular Blockade on Intra-Operative Blood Loss During Spinal Surgery, Randomized Double Blinded Clinical Trial
Brief Title: Comparison Of Deep Versus Moderate Neuromuscular Blockade on Intra-Operative Blood Loss During Spinal Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Refaat Shaaban Abd El-aal, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: spine surgery anesthesia
Record Dates: First submitted 2021-12-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Spine Fracture
Keywords: spine; surgery; anesthesia; blood loss
MeSH Terms: conditions — Spinal Fractures; Hemorrhage | interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: randomized double blinded clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep neuromuscular blockade (Active Comparator)
  Interventions: Drug: Rocuronium; Device: nerve stimulator
- moderate neuromuscular blockade (Active Comparator)
  Interventions: Drug: Rocuronium; Device: nerve stimulator

INTERVENTIONS:
Drug: Rocuronium — After applying standard monitoring of pulse oximetry, ECG, noninvasive blood pressure, general anesthesia will be induced with fentanyl 1 µg/kg and propofol 2-3 mg/kg and Rocuronium 0.6 mg/kg will be administered for muscle relaxation after loss of consciousness, under the guidance of neuromuscular blockade monitoring. Tracheal intubation will be performed at a train-of-four count of 0. After that end-tidal carbon dioxide and temperature will be continuously monitored during the procedure. Mechanical ventilation will be instituted with o2:air of 4 L/min, tidal volume of 6-8 ml/kg and respiratory rate appropriate to achieving end-tidal carbon dioxide of 30-35 mmHg. no positive end-expiratory pressure; and inspiratory/expiratory ratio 1: 2. The patient's position will then be changed from supine to prone. Ephedrine 4 mg (if mean arterial pressure < 60 mmHg and heart rate < 40 bpm), or atropine 0.5 to 1.0 mg (if heart rate < 40 bpm) are used to prevent hypotension or bradycardia
Device: nerve stimulator — Neuromuscular blockade monitoring will be established and continuously monitored after induction using the Train Of Four (TOF) at the adductor pollicis muscle on the opposite hand and wrist to radial artery cannulation. Two surface electrocardiography electrodes will be placed on cleaned skin overlying the ulnar nerve, with one electrode positioned on the ulnar side of the flexor carpi radialis tendon and the other positioned 3cm proximal to the first. The transducer is then positioned with the flat side against the thumb. Supramaximal stimuli will be applied after autonomic calibration of acceleromyograph after an initial tetanic stimulus. After confirming a train-of-four ratio of 95 to 105%, neuromuscular blockade monitoring will start. The train-of-four mode of supramaximal stimulation (0.2 ms duration, frequency 2 Hz, two s duration) will be applied at 15 s intervals, which last until the end of anaesthesia.

SUMMARY:
Reduction of intra-operative blood loss

DETAILED DESCRIPTION:
Spine surgery is usually performed using a posterior approach with the patient in the prone position, but on the other hand this position causes venous engorgement in the back and increases bleeding with the risk of interruption of surgery and increases the need for blood transfusion. The prone position also produces undesirable haemodynamic changes resulting from compression of large vessels and decreased venous return to the heart.

Deep neuromuscular blockade has been shown to improve surgical conditions compared with moderate neuromuscular blockade in various surgical procedures specially different laparoscopic procedures to optimize surgical field conditions. In spine surgery, although many other factors such as the body habitus of the patient and the surgical equipment are important, an improvement in surgical field conditions can be achieved through reducing muscle tension in the back, and also reducing intra-abdominal and thoracic pressure. This goal may be attainable by using deep neuromuscular blockade. Better operating conditions offer the surgeon easier access to the surgical field with less damage. However, the effect of deep neuromuscular blockade on surgical bleeding in spinal surgery in the prone position has been yet under evaluation.

The investigators hypothesise that deep, compared with moderate, neuromuscular blockade would cause less surgical bleeding in spinal surgery in the prone position. The investigators aim to evaluate the effects and superiority of deep neuromuscular blockade on surgical bleeding in patients undergoing posterior lumbar interbody fusion surgery in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years.
* American Society of Anesthesiologists physical status classification (ASA) I - III
* Patients scheduled for posterior lumbar interbody fusion (2-level or 3-level).

Exclusion Criteria:

* Urgent or emergency case or re-operation.
* History of pre-operative anticoagulant medication or an indication for peri-operative anticoagulant medication.
* ASA classification more than III.
* Age less than 16 years.
* Reduced left and right ventricular function (ejection fraction <40%).
* Previous respiratory disease or a diagnosed neuromuscular disorder.
* Pre-operative dysrhythmia.
* Allergy to neuromuscular blocking agents.
* Family history of malignant hyperthermia.
* Decreased renal function (serum creatinine level more than twice the normal range, urine output <0.5 ml kg/h, glomerular filtration ratio <60 ml/ h).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Volume of surgical bleeding. | Baseline
  Volume of surgical bleeding will be recorded before surgical field lavage, and again at the end of surgery, by measuring the total volume of blood collected in the suction bottle minus the lavage fluid volume used for wound irrigation.

SECONDARY OUTCOMES:
surgeon's satisfaction with the operating conditions | Baseline
  The score for the surgeon's satisfaction (lowest, 1; highest, 5) with the surgical conditions will be assessed at the end of surgery. Extremely poor (Score 1) indicated that the surgeon is unable to work because of an inability to obtain a visible field due to inadequate muscle relaxation; poor (Score 2) indicated that there is a visible field, but the surgeon is severely hampered by inadequate muscle relaxation; acceptable (Score 3) indicated that there is a wide visible field and acceptable muscle relaxation; good (Score 4) indicated a wide working field with adequate muscle relaxation; excellent (Score 5) indicated a wide visible working field without any muscle rigidity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Moneim Bakr Eid, Professor, Study Chair — 1.2; Ola Mahmoud Wahba Gnedy, Professor, Study Director — 1.1, 2.2, 3.4; Shimaa Abbas Hassan, Dr, Study Director — 1.3, 2.1

REFERENCES:
- [Background] Hatada T, Kusunoki M, Sakiyama T, Sakanoue Y, Yamamura T, Okutani R, Kono K, Ishida H, Utsunomiya J. Hemodynamics in the prone jackknife position during surgery. Am J Surg. 1991 Jul;162(1):55-8. doi: 10.1016/0002-9610(91)90202-o. PMID 2063971
- [Background] Wadsworth R, Anderton JM, Vohra A. The effect of four different surgical prone positions on cardiovascular parameters in healthy volunteers. Anaesthesia. 1996 Sep;51(9):819-22. doi: 10.1111/j.1365-2044.1996.tb12608.x. PMID 8882241
- [Background] Yokoyama M, Ueda W, Hirakawa M, Yamamoto H. Hemodynamic effect of the prone position during anesthesia. Acta Anaesthesiol Scand. 1991 Nov;35(8):741-4. doi: 10.1111/j.1399-6576.1991.tb03382.x. PMID 1763593
- [Background] Edgcombe H, Carter K, Yarrow S. Anaesthesia in the prone position. Br J Anaesth. 2008 Feb;100(2):165-83. doi: 10.1093/bja/aem380. PMID 18211991
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Van Wijk RM, Watts RW, Ledowski T, Trochsler M, Moran JL, Arenas GW. Deep neuromuscular block reduces intra-abdominal pressure requirements during laparoscopic cholecystectomy: a prospective observational study. Acta Anaesthesiol Scand. 2015 Apr;59(4):434-40. doi: 10.1111/aas.12491. Epub 2015 Feb 13. PMID 25684372
- [Background] Kim MH, Lee KY, Lee KY, Min BS, Yoo YC. Maintaining Optimal Surgical Conditions With Low Insufflation Pressures is Possible With Deep Neuromuscular Blockade During Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-Blind, Parallel-Group Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2920. doi: 10.1097/MD.0000000000002920. PMID 26945393
- [Background] Kang WS, Oh CS, Rhee KY, Kang MH, Kim TH, Lee SH, Kim SH. Deep neuromuscular blockade during spinal surgery reduces intra-operative blood loss: A randomised clinical trial. Eur J Anaesthesiol. 2020 Mar;37(3):187-195. doi: 10.1097/EJA.0000000000001135. PMID 31860601